CLINICAL TRIAL: NCT03406780
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of Intravenous Delivery of Allogeneic Cardiosphere-Derived Cells in Subjects With Duchenne Muscular Dystrophy
Brief Title: A Study of CAP-1002 in Ambulatory and Non-Ambulatory Patients With Duchenne Muscular Dystrophy
Acronym: HOPE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-1002-DMD-02
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Disorders, Atrophic; Muscular Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn
Keywords: Duchenne Muscular Dystrophy; Cell Therapy; Performance of the Upper Limb; Pulmonary Function; Ambulatory; Non-Ambulatory; Glucocorticoids
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Disorders, Atrophic; Muscular Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, X-Linked; Genetic Diseases, Inborn | interventions — chenodeoxycholate sulfate conjugate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAP-1002 (Experimental): Patients will receive 150 million Cardiosphere-derived Cells (CDCs) via intravenous infusion every 3 months for a total of 4 doses.
  Interventions: Biological: CAP-1002
- Placebo (Placebo Comparator): Patients will receive a placebo solution via intravenous infusion every 3 months for a total of 4 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CAP-1002 — The active pharmaceutical ingredient in CAP-1002 is Cardiosphere-Derived Cells (CDCs). CDCs are known to secrete numerous bioactive elements (growth factors, exosomes) which impact the therapeutic benefits of the cell-based therapy. The mechanism of action is the composite ability to be immunomodulatory, anti-fibrotic, anti-inflammatory, and pro-angiogenic.
  Other Names: Cardiosphere-Derived Cells; CDCs; deramiocel
  Arms: CAP-1002
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
HOPE-2 is a double-blind clinical trial evaluating the safety and efficacy of a cell therapy called CAP-1002 in study participants with Duchenne Muscular Dystrophy (DMD). Non-ambulatory and ambulatory boys and young men who meet eligibility criteria will be randomly assigned to receive either CAP-1002 or placebo every 3 months for a total of 4 doses during a 12-month period.

DETAILED DESCRIPTION:
* Approximately 20 eligible study participants will be randomized to either CAP-1002 or placebo in a 1:1 ratio.
* The trial will include visits at Screening, Baseline/Day 1, Week 4, and Months 3, 6, 9, and 12 with IV infusions of CAP-1002 or placebo on Day 1 and Months 3, 6, and 9.
* Safety evaluations will include adverse events, concomitant medications, physical exam, vital signs, 12-lead ECG, and clinical laboratory testing.
* Efficacy will be evaluated by Performance of the Upper Limb, cardiac MRI, pulmonary function testing, North Star Ambulatory Assessment (ambulatory subjects only), strength testing, and quality of life.
* If trial data suggests an appropriate risk/benefit profile of CAP-1002, Capricor, upon the recommendation of the Data Safety Monitoring Board (DSMB), will introduce an open-label extension study to offer CAP-1002 to study participants who were randomized to placebo and completed all trial visits during the 12-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants at least 10 years of age at time of consent
2. Participants willing and able to provide informed consent to participate in the trial if >= 18 years of age, and assent with parental or guardian informed consent if < 18 years of age
3. Participants with diagnosis of DMD based on clinical and phenotypic manifestations consistent with DMD (e.g., family history of DMD, elevated creatine kinase, dystrophin muscle biopsy, calf pseudohypertrophy, Gowers' sign, and gait impairment before 7 years of age) with confirmatory genetic testing performed at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
4. Participants with performance of the Upper Limb entry item score 2-5
5. Participants if ambulatory, 10-meter walk/run velocity < 1 meter/second
6. Participants with loss of independent ambulation by 18th birthday (standing unassisted or ability to take, at most, several steps independently is not considered ambulation)
7. Participants who receiving standard of care therapy at an experienced, multidisciplinary, DMD center as evidenced by regular cardiac and pulmonary monitoring, systemic glucocorticoid treatment, and at-home range of motion exercises
8. Participants who received treatment with a systemic glucocorticoid is required for at least 12 months prior to randomization. The dose must remain stable for at least 6 months prior to randomization with the exception of either weight-based dose adjustment or a decrease in steroid dose of ≤ 10% for toxicity. For patients on chronic deflazacort, treatment with an equivalent dose of prednisone or prednisolone for a period of ≤ 30 days to bridge lack of availability of deflazacort during the 6 months prior to randomization is acceptable
9. Participants with current and up-to-date immunizations according to children and adolescent Centers for Disease Control immunization schedule, unless contraindicated, including the following: meningococcal and meningococcal B; tetanus, diphtheria & acellular pertussis (Tdap); and pneumococcal polysaccharide vaccinations
10. Participants with adequate venous access for parenteral IP infusions and routine blood collections in the judgement of the Investigator
11. Participants assessed by the Investigator as willing and able to comply with the requirements of the trial

Exclusion Criteria:

1. Participants with Left Ventricular Ejection Fraction (LVEF) < 35%
2. Participants with elbow-flexion contractures > 30° in both extremities
3. Participants with Body Mass Index (BMI) > 45
4. Participants with documentation of exon 44 skip-amenable mutation(s) in the dystrophin gene
5. Participants with documentation of dystrophin deletion mutation(s) encompassing and limited to exons 3-7
6. Participants with percent predicted FVC (FVC%p) < 35%
7. Participants with inability to perform consistent FVC measurement within ±15% during paired testing at screening
8. Participants with risk of near-term respiratory decompensation in the judgment of the investigator, or the need for initiation of non-invasive ventilator support as defined by serum bicarbonate ≥ 29 mmol/L at screening
9. Participants with history of non DMD-related chronic respiratory disease requiring ongoing or intermittent treatment, including, but not limited to, asthma, bronchitis, and tuberculosis
10. Participants with acute respiratory illness within 30 days prior to screening
11. Participants with initiation of non-invasive ventilation within 30 days prior to screening, or the anticipated need to initiate non-invasive ventilation within the 12 months following screening
12. Participants with planned or anticipated thoracic or spinal surgery within the 12 months following randomization
13. Participants with planned or anticipated lower extremity surgery within the 12 months following randomization, if ambulatory
14. Participants with known hypersensitivity to Dimethyl Sulfoxide (DMSO) or bovine products
15. Participants with initiation of treatment with metformin or insulin within 3 months prior to randomization
16. Participants with initiation of treatment with an FDA-approved exon skipping therapy for the treatment of DMD within 24 months prior to randomization or dose adjustments to the therapy within 12 months prior to randomization with the exception of weight-based dose adjustments.
17. Participants who received treatment with Human Growth Hormone (HGH) within 3 months prior to randomization, unless on a stable dose (as determined by the site PI) for at least 24 months prior to randomization
18. Participants who received Treatment with idebenone within 3 months prior to randomization
19. Participants who received treatment with a cell therapy product within 12 months prior to randomization
20. Participants who received treatment with an investigational product within 6 months prior to randomization
21. Participants with history, or current use, of drugs or alcohol that could impair their ability to comply with participation in the trial
22. Participants with inability to comply with the investigational plan and follow-up visit schedule for any reason, in the judgment of the investigator

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig McDonald, MD, Principal Investigator — University of California, Davis
Locations (9):
- United States (9):
  - University of California, Davis, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDonald CM, Marban E, Hendrix S, Hogan N, Ruckdeschel Smith R, Eagle M, Finkel RS, Tian C, Janas J, Harmelink MM, Varadhachary AS, Taylor MD, Hor KN, Mayer OH, Henricson EK, Furlong P, Ascheim DD, Rogy S, Williams P, Marban L; HOPE-2 Study Group. Repeated intravenous cardiosphere-derived cell therapy in late-stage Duchenne muscular dystrophy (HOPE-2): a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2022 Mar 12;399(10329):1049-1058. doi: 10.1016/S0140-6736(22)00012-5. PMID 35279258
- See also: Company website — http://capricor.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 7 investigational sites in the United States from 04 April 2018 to 10 March 2020.
Pre-assignment Details: A total of 26 participants were screened, of these, 6 participants were deemed screen failures. Overall, 20 participants were randomized to receive CAP-1002 or placebo in this study.
Groups:
- CAP-1002: Participants received CAP-1002 at a dose of 150 million Cardiosphere-Derived Cells (CDCs) via intravenous infusion, every 3 months on Day 1 and at Months 3, 6, and 9.
- Placebo: Participants received a CAP-1002 matching placebo via intravenous infusion, every 3 months on Day 1 and at Months 3, 6, and 9.
Period: Overall Study
Arm/Group | CAP-1002 | Placebo
Started | 8 | 12
Treated | 8 | 12
Completed | 7 | 9
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAP-1002 | Placebo | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (3.44) | 14.4 (3.03) | 14.3 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 6 | 12 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Capacity as Assessed by the Mid-level (Elbow) Dimension Score of the Performance of Upper Limb (PUL) Version 1.2 at Month 12
Description: Change from baseline in functional capacity as assessed by the mid-level (elbow) dimension of PUL version 1.2 at Month 12 expressed as percentile ranked change.
  PUL 1.2 scale assesses motor performance in the upper limb. PUL 1.2 included 22 items. One entry item to define the starting functional level, and 21 items subdivided into: Shoulder Level (score 0 to 16); Elbow Level (score 0 to 34); Distal Level Dimension (score 0 to 24). The total score range was from 0 to 74. For all items, the higher the score, the better the outcome. A negative change indicates worst the outcome. Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Baseline, Month 12
Population: ITT population included participants who were randomized. Here, "overall number of participants" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank | 65.5 (10.82) | 29.3 (9.23)

2. Primary Outcome: Number of Participants Experiencing Acute Respiratory Decompensation
Description: Acute respiratory decompensation was defined as an unexplained rapid deterioration of the participant's condition with increasing shortness of breath requiring oxygen supplementation.
Time Frame: Baseline through Month 12
Population: ITT population included participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Hypersensitivity Reactions
Description: Hypersensitivity reaction was defined as a clinical syndrome including, but not limited to, fever, leukocytosis, or rash with onset less than or equal to (<=) 2 hours post-infusion and lasting less than (<) 24 hours, in the absence of clinical signs of concomitant infection.
Time Frame: Baseline through Month 12
Population: ITT population included participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Participants | 3 | 0

4. Primary Outcome: Number of Participants With All-cause Mortality
Description: Number of participants who died due to any cause were reported.
Time Frame: Baseline through Month 12
Population: Safety population included all participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE was defined as an AE that results in any of the following outcomes: Death; life-threatening adverse event; Inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; congenital anomaly/birth defect.
Time Frame: Baseline through Month 12
Population: Safety population included all participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Participants | 2 | 0

6. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Related to Investigational Product (IP) or Administration Procedure
Description: TEAE was defined as an AE that was not present prior to the initiation of line placement procedure for the IP infusion or was present but worsened in intensity or frequency. The Investigator assessed the relationship (causality) of an AE to the investigational product and administration procedure.
Time Frame: Baseline through Month 12
Population: Safety population included all participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Participants | 5 | 5

7. Primary Outcome: Number of Participants With Immune Sensitization Syndrome
Description: Immune sensitization syndrome is defined as a) clinical signs and symptoms that are consistent with systemic inflammation (e.g.,fever, leukocytosis, rash, arthralgia), with an onset >=24 hours after infusion of the investigational product, in the absence of clinical signs of concomitant infection, and b) an elevation of anti-Human Leukocyte Antigen (anti-HLA) antibodies against the Donor-Specific Antibody (DSA) cells, which is detected <=30 days after the onset of syndrome, that meets the following criteria: i) 2000 mean fluorescence intensity if mean fluorescence intensity is <=1000 at baseline, or ii) >=2 times the baseline value.
Time Frame: Baseline through Month 12
Population: Safety population included all participants who received investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With TEAEs and Severity of TEAEs
Description: TEAE was defined as an AE that was not present prior to the initiation of line placement procedure for the IP infusion or was present but worsened in intensity or frequency. Severity of TEAEs were determined by following criteria:: Mild (Grade 1): Transient or mild discomfort; no limitation in activity; no medical intervention/therapy required; Moderate (Grade 2): Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required; Severe (Grade 3): Marked limitation in activity, some assistance usually required; medical intervention/therapy required and often requiring hospitalization or prolongation of hospitalization; Life-Threatening or Disabling (Grade 4): Extreme limitation in activity, significant assistance required; significant medical intervention/therapy required; hospitalization, prolongation of hospitalization, or hospice care; Fatal (Grade 5): death.
Time Frame: Baseline through Month 12
Population: Safety population included all participants who received investigational product. Here, "overall number of participants" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
participants
  Participants with TEAEs | 7 | 12
  Participants with Mild (Grade 1) TEAEs | 1 | 6
  Participants with Moderate (Grade 2) TEAEs | 4 | 5
  Participants with Severe (Grade 3) TEAEs | 1 | 1
  Participants with Life-threatening or Disabling (Grade 4) TEAEs | 1 | 0
  Participants with Fatal (Grade 5) TEAEs | 0 | 0

9. Secondary Outcome: Change From Baseline in the Mid-level (Elbow) Dimension Score of the PUL 1.2 at Months 3, 6, and 9
Description: Change From Baseline in the Mid-level (Elbow) Dimension Score of the PUL 1.2 at Months 3, 6, and 9 expressed as percentile ranked change.
  PUL 1.2 scale assesses motor performance in the upper limb. PUL 1.2 included 22 items. One entry item to define the starting functional level, and 21 items subdivided into: Shoulder Level (score 0 to 16); Elbow Level (score 0 to 34); Distal Level Dimension (score 0 to 24). The total score range was from 0 to 74. For all items, the higher the score, the better the outcome. A negative change indicates worst the outcome. Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Baseline, Months 3, 6, and 9
Population: ITT population included participants who were randomized. Here, "overall number of participants" signifies those participants who were evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for specified time points.
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  At Month 3 | 86.6 (10.51) | 66.8 (8.40)
  At Month 6 | 77.6 (11.19) | 49.9 (8.38)
  At Month 9 | 68.1 (10.83) | 48.4 (8.97)

10. Secondary Outcome: Change From Baseline in Regional Systolic Left Ventricular (LV) Wall Thickening, as Assessed by Cardiac Magnetic Resonance Imaging (MRI) at Months 6 and 12
Description: Change from baseline in regional systolic LV wall thickening (anterior, lateral, inferior, septal) expressed as percentile ranked change, as assessed by cardiac MRI at Months 6 and 12.
  Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  Systolic Wall Thickening Anterior LV at Month 6 | 46.3 (10.84) | 45.8 (7.13)
  Systolic Wall Thickening Anterior LV at Month 12 | 40.9 (8.90) | 40.7 (8.88)
  Systolic Wall Thickening Lateral LV at Month 6 | 50.4 (18.47) | 39.9 (12.32)
  Systolic Wall Thickening Lateral LV at Month 12 | 49.2 (17.00) | 27.4 (14.26)
  Systolic Wall Thickening Inferior LV at Month 6 | 57.3 (12.37) | 59.7 (8.52)
  Systolic Wall Thickening Inferior LV at Month 12 | 60.3 (10.99) | 45.7 (9.94)
  Systolic Wall Thickening Septal LV at Month 6 | 50.1 (16.89) | 49.2 (11.34)
  Systolic Wall Thickening Septal LV at Month 12 | 50.8 (15.28) | 49.9 (12.97)

11. Other Pre Specified Outcome: Change From Baseline in Left Ventricular Ejection Fraction at Month 6 and 12
Description: Change from baseline in Left Ventricular Ejection Fraction assessed by cardiac magnetic resonance imaging (MRI) and expressed as percentile ranked change.
  Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Month 6 and 12
Population: Intent-to-Treat (ITT) Population includes all participants who are randomized. Participants were summarized and analyzed in the treatment group to which they were randomized. Number analyzed signifies participants evaluable for specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  Month 6 | 57.9 (11.00) | 34.9 (7.46)
  Month 12 | 54.5 (9.08) | 8.9 (9.29)

12. Other Pre Specified Outcome: Change From Baseline in Left Ventricular End-diastolic Volume at Month 6 and 12
Description: Change from baseline in Left Ventricular End-diastolic Volume assessed by cardiac magnetic resonance imaging (MRI) expressed as percentile ranked change.
  Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Month 6 and 12
Population: The ITT population includes all participants who are randomized. Participants were summarized and analyzed in the treatment group to which they were randomized. Number analyzed signifies participants evaluable for specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  Month 6 | 54.7 (12.89) | 33.4 (8.87)
  Month 12 | 49.2 (12.55) | 48.6 (11.81)

13. Other Pre Specified Outcome: Change From Baseline in Left Ventricular End-Diastolic Volume (Indexed) at Month 6 and 12
Description: Change from baseline in Left Ventricular End-diastolic Volume (Indexed) assessed by cardiac magnetic resonance imaging (MRI) expressed as percentile ranked change.
  The End-diastolic Volume (Indexed) (EDVI) is calculated as follows: EDVI= EDV (End-diastolic Volume)/BSA (body surface area) = xxx mL/m^2. Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Month 6 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  Month 6 | 34.8 (14.11) | 58.1 (11.51)
  Month 12 | 12.2 (13.29) | 60.0 (12.27)

14. Other Pre Specified Outcome: Change From Baseline in Left Ventricular End-Systolic Volume at Month 6 and 12
Description: Change from baseline in Left Ventricular End-systolic Volume assessed by cardiac magnetic resonance imaging (MRI) expressed as percentile ranked change.
  Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Month 6 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  Month 6 | 48.4 (12.16) | 51.1 (8.44)
  Month 12 | 33.3 (10.97) | 79.2 (10.52)

15. Other Pre Specified Outcome: Change From Baseline in Left Ventricular End-Systolic Volume (Indexed) at Month 6 and 12
Description: Change from baseline in Left Ventricular End-systolic Volume (Indexed) assessed by cardiac magnetic resonance imaging (MRI) expressed as percentile ranked change.
  The End-systolic Volume (Indexed) (ESVI) is calculated as follows: ESVI= ESV (End-systolic Volume)/BSA (body surface area) = xxx mL/m^2. Change from baseline and baseline values were converted to a percentile rank over all timepoints and at baseline using a non-parametric version of the prespecified model, generated by calculating the percentile rank of each change-from-baseline value relative to all observed change-from-baseline values for the same outcome (across all patients and all post-baseline observation times).
Time Frame: Month 6 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Percentile Rank
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 8 | 12
Percentile Rank
  Month 6 | 38.6 (12.96) | 50.2 (10.73)
  Month 12 | 15.8 (12.27) | 68.9 (11.77)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: Safety population included all participants who received investigational product.
Arm/Group | CAP-1002 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/12
Other Adverse Events (participants affected / at risk) | 7/8 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAP-1002 (N=8) | Placebo (N=12)
Allergic Reaction To Excipient (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAP-1002 (N=8) | Placebo (N=12)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 1 (1)
Myopia (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Tooth Impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Vessel Puncture Site Haematoma (General disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 4 (5)
Otitis Media Acute (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fracture Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Compression Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT03406780/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03406780/SAP_002.pdf